CLINICAL TRIAL: NCT01118390
Title: Treatment of Leg Telangiectasias With Nd:YAG 1064nm
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Grupo de Cirurgia Vascular (Other)
Responsible Party: Marco Antonio Munia, Departamento de Cirurgia Vascular HCFMUSP
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0072/09
Record Dates: First submitted 2010-04-29; First posted 2010-05-06 (Estimated); Last update posted 2010-05-06 (Estimated); Status verified 2009-08

CONDITIONS: Telangiectasias
Keywords: telangiectasias; leg; sclerotherapy; laser; glycose
MeSH Terms: conditions — Telangiectasis | interventions — Lasers; Sclerotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laser Nd:YAG 1064nm (Experimental): Patients with leg telangiectasias are treated with 3 sessions of Nd:YAG 1064nm, with 14 days interval
  Interventions: Device: Laser Nd:YAG 1064nm
- Sclerotherapy (Active Comparator): Patients with leg telangiectasias are treated with 3 sessions of sclerotherapy, with 14 days interval
  Interventions: Other: Sclerotherapy

INTERVENTIONS:
Device: Laser Nd:YAG 1064nm — Patients with leg telangiectasias are treated with 3 sessions of Nd:YAG 1064nm, with 14 days interval
  Other Names: laser; Xeo; Cool Glide
  Arms: Laser Nd:YAG 1064nm
Other: Sclerotherapy — Patients with leg telangiectasias are treated with 3 sessions of sclerotherapy, with 14 days interval
  Other Names: glicose
  Arms: Sclerotherapy

SUMMARY:
Studying the results of treatment of dilated vessels of the lower limbs with laser, and compare them to those obtained with sclerotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with leg telangiectasias

Exclusion Criteria:

* Arterial disease
* Varices
* Diabetes

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-08; Primary Completion 2010-03 (Actual); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
treatment of leg telangiectasias | first day
  Patients respond after treatment a questionnaire about satisfaction for both the laser and for conventional sclerotherapy.
Treatment of telangiectasias | 1 month
  Patients respond after treatment a questionnaire about satisfaction for both the laser and for conventional sclerotherapy.

SECONDARY OUTCOMES:
Presence of adverse effects | after 1 month
  Patients are monitored to adverse effects such as blemishes, scars and ulcers
Pain Scores on the Visual Analog Scale | After 1 month
  Patients evaluate pain on the Visual Analog Scale

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Wolosker, MD, PhD, Study Chair — Hospital das Clinicas, University of Sao Paulo; Marco Munia, MD, Principal Investigator — Hospital das Clinicas, University of Sao Paulo
Locations (1):
- Hospital das Clinicas da FMUSP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Anderson RR, Parrish JA. Selective photothermolysis: precise microsurgery by selective absorption of pulsed radiation. Science. 1983 Apr 29;220(4596):524-7. doi: 10.1126/science.6836297.
- [Background] Coles CM, Werner RS, Zelickson BD. Comparative pilot study evaluating the treatment of leg veins with a long pulse ND:YAG laser and sclerotherapy. Lasers Surg Med. 2002;30(2):154-9. doi: 10.1002/lsm.10028. PMID 11870796
- [Background] Baumler W, Ulrich H, Hartl A, Landthaler M, Shafirstein G. Optimal parameters for the treatment of leg veins using Nd:YAG lasers at 1064 nm. Br J Dermatol. 2006 Aug;155(2):364-71. doi: 10.1111/j.1365-2133.2006.07314.x. PMID 16882176
- [Background] Dudelzak J, Hussain M, Goldberg DJ. Vascular-specific laser wavelength for the treatment of facial telangiectasias. J Drugs Dermatol. 2009 Mar;8(3):227-9. PMID 19271368